CLINICAL TRIAL: NCT03912246
Title: Collection d'échantillons Biologiques Humains de Sujets Sains et Malades Pour la Mise au Point et la Validation de Nouvelles méthodes de Diagnostic et Pour la réalisation d'Expertises Dans le Domaine Des Maladies Infectieuses et Tropicales
Brief Title: Collection of Human Biological Samples for the Development and Validation of New Methods of Diagnosis and for the Realization of Expertises Diagnostics in the Field of Infectious Diseases and Tropical
Acronym: Diagmicoll
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2008-16; DC-2008-68 (Other: Institut Pasteur)
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Infectious Disease; Tropical Disease
Keywords: sample; diagnostic
MeSH Terms: conditions — Communicable Diseases; Disease | interventions — Spinal Puncture

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Healthy volunteers (Experimental): Human biological samples:
  whole blood (serum or plasma, PBMCs, red blood cells), urine, feces, saliva, tears, mouth and skin swabs.
  Bio-clinical data :
  adjusted to the purpose of the searches will be collected
  Interventions: Biological: biological samples
- Patients with neuro-meningeal infection (Experimental): Human biological samples:
  Whole blood (serum or plasma, PBMCs, red blood cells), urine, feces, saliva, tears, mouth and skin swabs.
  Extended collection of CSF
  Bio-clinical data :
  adjusted to the purpose of the searches will be collected
  Interventions: Biological: biological samples; Procedure: lumbar puncture

INTERVENTIONS:
Biological: biological samples — collection of blood, urine, saliva, stool, skin and mouth swabs, tears
Procedure: lumbar puncture — collection of cerebrospinal fluid
  Arms: Patients with neuro-meningeal infection

SUMMARY:
Direct constitution of collections from various samples taken on a prospective cohort of healthy volunteers, to prepare human biological samples of known characteristics (biochemical and serological in particular) and quality controlled.

DETAILED DESCRIPTION:
Direct constitution of collection from various samples taken on a prospective cohort of healthy volunteers, to prepare human biological samples of known characteristics (biochemical and serological in particular) and quality controlled.

This collection will allow, as a priority, a development stage, ie the establishment of the proof of concept of new diagnostic methods in the field of infectious and tropical diseases.

There will be 2 cohorts (= arms) for this study: the main cohort of healthy volunteers and the N cohort, which will consist of patients with neuro-meningeal disease of infectious appearance and followed in specialized consultation.

ELIGIBILITY:
Inclusion Criteria:

* major subject
* affiliated or benefiting from social security
* having signed the information and consent form
* negative HIV and HCV serology and negative HBV or vaccine serology (or old healed infection profile)
* for cohort N: neuromeningeal infection during dianostic exploration

Exclusion Criteria:

* Volunteers with a severe or chronic pathology significantly disturbing one or more bio-clinical parameters and / or requiring the regular intake of certain drugs (anti-inflammatories or corticosteroids for example).
* Woman whose pregnancy is known during the visit.
* Acute infection within 15 days or taking antiviral, antibiotic, antifungal or antiparasitic drugs in the last 15 days.
* Subject participating in a biomedical research or in a period of exclusion of a biomedical research.
* When monitoring O +, AB +, A + and B + blood group whose erythrocyte base is kept for CEPIA research, in case of antimalarial (travel), a minimum of 5 half-lives after the last dose of antimalaria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2009-04-27 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
development of new diagnostic methods | during all the study
  This collection will allow, as a priority, a first stage of development, that is to say the completion of the proof of concept of new diagnostic methods in the field of infectious and tropical diseases.

SECONDARY OUTCOMES:
performance improvement | during all the study
  In a second step, the collection will be able to improve the essential performances (sensitivity and specificity) of the methods to the study compared to the existing methods: speed, simplicity (molecular methods, etc) and cost; and may also uncover new non-infectious biomarkers.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre d'infectiologie, hopitale Necker, Paris
  - Institut Pasteur, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pajot A, Michel ML, Mancini-Bourgine M, Ungeheuer MN, Ojcius DM, Deng Q, Lemonnier FA, Lone YC. Identification of novel HLA-DR1-restricted epitopes from the hepatitis B virus envelope protein in mice expressing HLA-DR1 and vaccinated human subjects. Microbes Infect. 2006 Oct;8(12-13):2783-90. doi: 10.1016/j.micinf.2006.08.009. Epub 2006 Sep 12. PMID 17045504
- [Background] Buffet PA, Milon G, Brousse V, Correas JM, Dousset B, Couvelard A, Kianmanesh R, Farges O, Sauvanet A, Paye F, Ungeheuer MN, Ottone C, Khun H, Fiette L, Guigon G, Huerre M, Mercereau-Puijalon O, David PH. Ex vivo perfusion of human spleens maintains clearing and processing functions. Blood. 2006 May 1;107(9):3745-52. doi: 10.1182/blood-2005-10-4094. Epub 2005 Dec 29. PMID 16384927
- [Background] Launay O, Toneatti C, Bernede C, Njamkepo E, Petitprez K, Leblond A, Larnaudie S, Goujon C, Ungeheuer MN, Ajana F, Raccurt C, Beytout J, Chidiac C, Bouhour D, Guillemot D, Guiso N. Antibodies to tetanus, diphtheria and pertussis among healthy adults vaccinated according to the French vaccination recommendations. Hum Vaccin. 2009 May;5(5):341-6. doi: 10.4161/hv.5.5.7575. Epub 2009 May 9. PMID 19221513
- [Background] Taneja N, Nato F, Dartevelle S, Sire JM, Garin B, Thi Phuong LN, Diep TT, Shako JC, Bimet F, Filliol I, Muyembe JJ, Ungeheuer MN, Ottone C, Sansonetti P, Germani Y. Dipstick test for rapid diagnosis of Shigella dysenteriae 1 in bacterial cultures and its potential use on stool samples. PLoS One. 2011;6(10):e24830. doi: 10.1371/journal.pone.0024830. Epub 2011 Oct 3. PMID 21984895
- [Background] Azimi-Nezhad M, Lambert D, Ottone C, Perrin C, Chapel C, Gaillard G, Pfister M, Masson C, Tabone E, Betsou F, Meyronet D, Ungeheuer MN, Siest SV. Influence of pre-analytical variables on VEGF gene expression and circulating protein concentrations. Biopreserv Biobank. 2012 Oct;10(5):454-61. doi: 10.1089/bio.2012.0016. PMID 24845047
- [Background] Berthet N, Paulous S, Coffey LL, Frenkiel MP, Moltini I, Tran C, Matheus S, Ottone C, Ungeheuer MN, Renaudat C, Caro V, Dussart P, Gessain A, Despres P. Resequencing microarray method for molecular diagnosis of human arboviral diseases. J Clin Virol. 2013 Mar;56(3):238-43. doi: 10.1016/j.jcv.2012.10.022. Epub 2012 Dec 7. PMID 23219893
- [Background] Duran C, Nato F, Dartevelle S, Thi Phuong LN, Taneja N, Ungeheuer MN, Soza G, Anderson L, Benadof D, Zamorano A, Diep TT, Nguyen TQ, Nguyen VH, Ottone C, Begaud E, Pahil S, Prado V, Sansonetti P, Germani Y. Rapid diagnosis of diarrhea caused by Shigella sonnei using dipsticks; comparison of rectal swabs, direct stool and stool culture. PLoS One. 2013 Nov 22;8(11):e80267. doi: 10.1371/journal.pone.0080267. eCollection 2013. PMID 24278267
- [Background] Fremond ML, Perot P, Muth E, Cros G, Dumarest M, Mahlaoui N, Seilhean D, Desguerre I, Hebert C, Corre-Catelin N, Neven B, Lecuit M, Blanche S, Picard C, Eloit M. Next-Generation Sequencing for Diagnosis and Tailored Therapy: A Case Report of Astrovirus-Associated Progressive Encephalitis. J Pediatric Infect Dis Soc. 2015 Sep;4(3):e53-7. doi: 10.1093/jpids/piv040. Epub 2015 Jul 12. PMID 26407445
- [Background] Vayssier-Taussat M, Cosson JF, Degeilh B, Eloit M, Fontanet A, Moutailler S, Raoult D, Sellal E, Ungeheuer MN, Zylbermann P. How a multidisciplinary 'One Health' approach can combat the tick-borne pathogen threat in Europe. Future Microbiol. 2015;10(5):809-18. doi: 10.2217/fmb.15.15. PMID 26000651
- [Background] Neven B, Perot P, Bruneau J, Pasquet M, Ramirez M, Diana JS, Luzi S, Corre-Catelin N, Chardot C, Moshous D, Leclerc Mercier S, Mahlaoui N, Aladjidi N, Le Bail B, Lecuit M, Bodemer C, Molina TJ, Blanche S, Eloit M. Cutaneous and Visceral Chronic Granulomatous Disease Triggered by a Rubella Virus Vaccine Strain in Children With Primary Immunodeficiencies. Clin Infect Dis. 2017 Jan 1;64(1):83-86. doi: 10.1093/cid/ciw675. Epub 2016 Oct 6. PMID 27810866
- [Background] Guet-Revillet H, Jais JP, Ungeheuer MN, Coignard-Biehler H, Duchatelet S, Delage M, Lam T, Hovnanian A, Lortholary O, Nassif X, Nassif A, Join-Lambert O. The Microbiological Landscape of Anaerobic Infections in Hidradenitis Suppurativa: A Prospective Metagenomic Study. Clin Infect Dis. 2017 Jul 15;65(2):282-291. doi: 10.1093/cid/cix285. PMID 28379372
- [Background] Charlier C, Perrodeau E, Leclercq A, Cazenave B, Pilmis B, Henry B, Lopes A, Maury MM, Moura A, Goffinet F, Dieye HB, Thouvenot P, Ungeheuer MN, Tourdjman M, Goulet V, de Valk H, Lortholary O, Ravaud P, Lecuit M; MONALISA study group. Clinical features and prognostic factors of listeriosis: the MONALISA national prospective cohort study. Lancet Infect Dis. 2017 May;17(5):510-519. doi: 10.1016/S1473-3099(16)30521-7. Epub 2017 Jan 28. PMID 28139432
- [Background] Belizna C, Stojanovich L, Cohen-Tervaert JW, Fassot C, Henrion D, Loufrani L, Nagy G, Muchardt C, Hasan M, Ungeheuer MN, Arnaud L, Alijotas-Reig J, Esteve-Valverde E, Nicoletti F, Saulnier P, Godon A, Reynier P, Chretien JM, Damian L, Omarjee L, Mahe G, Pistorius MA, Meroni PL, Devreese K. Primary antiphospholipid syndrome and antiphospholipid syndrome associated to systemic lupus: Are they different entities? Autoimmun Rev. 2018 Aug;17(8):739-745. doi: 10.1016/j.autrev.2018.01.027. Epub 2018 Jun 6. PMID 29885541
- [Background] Belizna C, Pregnolato F, Abad S, Alijotas-Reig J, Amital H, Amoura Z, Andreoli L, Andres E, Aouba A, Apras Bilgen S, Arnaud L, Bienvenu B, Bitsadze V, Blanco P, Blank M, Borghi MO, Caligaro A, Candrea E, Canti V, Chiche L, Chretien JM, Cohen Tervaert JW, Damian L, Delross T, Dernis E, Devreese K, Djokovic A, Esteve-Valverde E, Favaro M, Fassot C, Ferrer-Oliveras R, Godon A, Hamidou M, Hasan M, Henrion D, Imbert B, Jeandel PY, Jeannin P, Jego P, Jourde-Chiche N, Khizroeva J, Lambotte O, Landron C, Latino JO, Lazaro E, de Leeuw K, Le Gallou T, Kilic L, Limper M, Loufrani L, Lubin R, Magy-Bertrand N, Mahe G, Makatsariya A, Martin T, Muchardt C, Nagy G, Omarjee L, Van Paasen P, Pernod G, Perrinet F, Pires Rosa G, Pistorius MA, Ruffatti A, Said F, Saulnier P, Sene D, Sentilhes L, Shovman O, Sibilia J, Sinescu C, Stanisavljevic N, Stojanovich L, Tam LS, Tincani A, Tollis F, Udry S, Ungeheuer MN, Versini M, Cervera R, Meroni PL. HIBISCUS: Hydroxychloroquine for the secondary prevention of thrombotic and obstetrical events in primary antiphospholipid syndrome. Autoimmun Rev. 2018 Dec;17(12):1153-1168. doi: 10.1016/j.autrev.2018.05.012. Epub 2018 Oct 12. PMID 30316994